CLINICAL TRIAL: NCT03371797
Title: Efficacy and Safety of Single Pill Combination (Amlodipine/Valsartan) in Hypertensive Patients Not Controlled on Previous Monotherapy: An Observational Real Life Study
Brief Title: Amlodipine VaLsartan Efficacy in Hypertensive Patients.A Real World Trial
Acronym: ALERT
Status: Completed | Type: Observational
Sponsor: PharmEvo Pvt Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PE/PK/ALERT/SP/2017-01
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2017-12

CONDITIONS: Essential Hypertension
Keywords: ALERT, MSSBP, MSDBP
MeSH Terms: conditions — Essential Hypertension | interventions — Amlodipine, Valsartan Drug Combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Valsartan, Amlodipine single pill combination.The recommended dosage of AVSAR (Valsartan/Amlodipine) is one tablet per day.
  Interventions: Drug: Valsartan, Amlodipine -

INTERVENTIONS:
Drug: Valsartan, Amlodipine - — Valsartan is a non-peptide, orally active, and specific angiotensin II receptor blocker acting on the AT1 receptor subtype used as an antihypertensive agent.
  Amlodipine besylate is a dihydropyridine long-acting calcium channel blocker.
  Other Names: AVSAR

SUMMARY:
To determine the efficacy of valsartan/amlodipine 80/5 mg once daily dose is reducing mean sitting systolic blood pressure (MSSBP) and mean sitting diastolic blood pressure (MSDBP) after 8 weeks of therapy.

DETAILED DESCRIPTION:
Avsar in tablet form which contains two antihypertensive compounds with complementary mechanisms to control blood pressure in patients with essential hypertension: amlodipine belongs to the calcium antagonist class and valsartan to the angiotensin II antagonist class of medicines Amlodipine is a dihydropyridine calcium channel blocker that inhibits the transmembrane influx of calcium ions into vascular smooth muscle and cardiac muscle. Amlodipine is a peripheral arterial vasodilator that acts directly on vascular smooth muscle to cause a reduction in peripheral vascular resistance and reduction in blood pressure.Valsartan blocks the vasoconstrictor and aldosterone-secreting effects of angiotensin II by selectively blocking the binding of angiotensin II to the AT1 receptor in many tissues, such as vascular smooth muscle and the adrenal gland International studies are available concerning the single pill combination therapy used in Blood pressure reduction. To determine the clinical significance of single pill combination, conducted multi center real life study i.e.; "ALERT Trial" in our local population. Through this study, observed the effect of single pill combination on BP reduction and adverse events in health care settings. Antihypertensive drugs use in a single pill combination may further enhance BP control by reducing pill burden and improve patient compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose BP is >139/89mmHg and on monotherapy with minimum last 30 days
* Male or female aged (18 years - 70 Years)
* Signed informed consent

Exclusion Criteria:

* Secondary Hypertension
* Pregnant or Lactating mother
* Hypersensitivity to any active ingredient
* Peripheral artery disease
* Hepatic disease or biliary tract obstruction
* Chronic kidney disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ages Eligible for Study: 18 years - 70 Years Genders Eligible for Study: Both
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of valsartan/amlodipine 80/5 mg once daily dose is reducing mean sitting systolic blood pressure (MSSBP) and mean sitting diastolic blood pressure after 8 weeks of therapy. | 8 weeks
  To determine the efficacy of valsartan/amlodipine 80/5 mg once daily dose is reducing mean sitting systolic blood pressure (MSSBP) after 8 weeks of therapy.
  [Designated as safety issue: No]

SECONDARY OUTCOMES:
Measure percentage of participant with blood pressure change of <139/89 mmHg at the end of 8 week | 8 weeks
  To measure percentage of participant with blood pressure change of <139/89 mmHg at the end of 8 week
  [Designated as safety issue: No]
Participants experiencing adverse effect after taking single pill combination | 8 weeks
  Proportion of participants experiencing adverse effect after taking single pill combination
  [Designated as safety issue: Yes]

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem Ahsan, MBBS, Principal Investigator — PharmEvo Pvt Ltd
Locations (1):
- Medicell, Karachi, Sindh, Pakistan